CLINICAL TRIAL: NCT05869695
Title: Transcultural Adaptation and Validation to Spanish of the Optimal Screening for Prediction of Referral and Outcome (OSPRO) Questionnaires for Review-Of-Systems (OSPRO-ROS) and Yellow-Flags (OSPRO-YF) in Subjects With Musculoskeletal Pain.
Brief Title: Transcultural Adaptation and Validation to Spanish of the OSPRO Questionnaires
Acronym: SpanishOSPRO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Valencia (Other)
Collaborators: University of Alcala (Other); Escoles Universitaries Gimbernat (Other); Hospital ASEPEYO Sant Cugat (Unknown); Consorci Sanitari de Terrassa (Other)
Responsible Party: Principal Investigator, Enrique Lluch Girbés, Associate Professor, University of Valencia
Other Study IDs: 102999
Record Dates: First submitted 2023-05-05; First posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Musculoskeletal Pain
Keywords: OSPRO; Review of Systems; Red Flags; Psychosocial factors; Yellow Flags; Cross-cultural; Reliability; Validity
MeSH Terms: conditions — Musculoskeletal Pain | interventions — Patient Health Questionnaire

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- OSPRO-ROS: 100 patients presenting musculoskeletal pain: Patients between 18 and 75 years of age with primary complaints involving the cervical spine, lumbar spine, shoulder or knee. Were able to read and comprehend Spanish.
  Interventions: Other: OSPRO-ROS Questionnaire
- OSPRO-YF: 100 patients presenting musculoskeletal pain: Patients between 18 and 75 years of age with primary complaints involving the cervical spine, lumbar spine, shoulder or knee. Were able to read and comprehend Spanish.
  Interventions: Other: OSPRO-YF Questionnaire

INTERVENTIONS:
Other: OSPRO-ROS Questionnaire — Completion of questionnaires
  Other Names: Result of complementary tests; OSPRO-ROS retest
  Groups: OSPRO-ROS: 100 patients presenting musculoskeletal pain
Other: OSPRO-YF Questionnaire — Completion of questionnaires
  Other Names: Chronic Pain Acceptance Questionnaire (CPAQ); Fear-Avoidance Beliefs Questionnaire (FABQ); Pain Catastrophizing Scale (PCS); Patient Health Questionnaire-9 (PHQ-9); State Trait Anxiety Inventory (STAI); Tampa Scale for Kinesiophobia-11 (TSK-11); OSPRO-YF retest
  Groups: OSPRO-YF: 100 patients presenting musculoskeletal pain

SUMMARY:
Clinical guidelines for managing musculoskeletal pain recommend first, assessing and identifying any signs of severe physical conditions (i.e."red flags") and then, asessing the psychosocial prognostic factors of poor outcomes (i.e."yellow flags"). The Optimal Sreening for Prediction of Referral and Outcome (OSPRO) cohort studies were designed to develop and validate standard assessment tools for Review Of Systems (OSPRO-ROS) and Yellow Flags (OSPRO-YF).

DETAILED DESCRIPTION:
The objectives of this study were to translate and cross-cultural adapt OSPRO-ROS and OSPRO-YF questionnaires to Spanish and to investigate their psychometric properties for their use in subjects with musculoskeletal pain.To accomplish the objectives proposed, this study was developed in two phases:Phase I: Cross-cultural adaptation process.Phase II: Psychometric properties evaluation.

ELIGIBILITY:
Inclusion Criteria:

OSPRO-ROS:

1. Were coming to the emergency department on their first visit.
2. With acute musculoskeletal pain.
3. Were able to read and comprehed Spanish language.

OSPRO-YF:

1. Were seeking outpatient physical therapy treatment.
2. With chronic musculoskeletal pain involving the cervical spine, lumbar spine, shoulder or knee.
3. Were able to read and comprehend Spanish language.

Exclusion Criteria:

1. Widespread chronic pain syndrome (e.g. fibromyalgia or irritable bowel syndrome).
2. Neuropathic pain syndrome (e.g. complex regional pain syndrome or diabetic neuropathy).
3. Psychiatric history (currently in care of mental health care provider or taking > 2 precription psychiatric medications)
4. Cancer (currently receiving treatment for active cancer)
5. Neurological disorder (e.g. stroke, spinal cord injury, or traumatic brain injury).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: OSPRO-ROS:
  Person between 18 and 75 years of age who goes to the emergency department, presenting acute musculoskeletal pain with primary complaints involving the cervical spine, lumbar spine, shoulder or knee.
  OSPRO-YF:
  Person between 18 and 75 years of age who goes to the rehabilitation department, presenting chronic musculoskeletal pain with primary complaints involving the cervical spine, lumbar spine, shoulder or knee.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-11-30 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Patient-Reported Outcome Measure (PROM) development: Translation and Cross Cultural Adaptation to the Spanish population of the Optimal Screening for Prediction of Referral and Outcome (OSPRO) questionnaires. | from September 2018 to July 2021
  Two native Spanish speakers, health experienced in musculoskeletal pain and knowledge of English, translated into Spanish the Optimal Screening for Prediction of Referral and Outcome-Review of Systems (OSPRO-ROS) questionnaire original (English) and the Optimal Screening for Prediction of Referral and Outcome Yellow-Flags (OSPRO-YF) original questionnaire (English).
  Two native English speakers, knowledge of Spanish, reverse-translate the text to Spanish.
  25 participants with musculoskeletal pain completed the Optimal Screening for Prediction of Referral and Outcome (OSPRO) questionnaires.
  This outcome will be evaluated according the Consensus-based Standards for the selections of health Measurement Instruments (COSMIN) Risk of Bias checklist for PROMs, using their scoring manual: very good/adequate/doubtful/inadequate/NA for each standar.

SECONDARY OUTCOMES:
OSPRO questionnaires Psychometric property Validation | from January to June 2024
  The validity and reliability of the Spanish version translated from the questionnaires Optimal Screening for Prediction of Referral and Outcome (OSPRO) will be assessed.
  This outcome will be evaluated according the Consensus-based Standards for the selections of health Measurement Instruments (COSMIN) Risk of Bias checklist for PROMs, using their scoring manual: very good/adequate/doubtful/inadequate/NA for each standar.

CONTACTS AND LOCATIONS:
Overall Officials: ENRIQUE LLUCH GIRBÉS, Principal Investigator — UNIVERSITAT DE VALÈNCIA
Locations (2):
- Spain (2):
  - Hospital Asepeyo Sant Cugat, Sant Cugat del Vallès, Barcelona
  - Consorci Sanitari de Terrassa, Terrassa, Barcelona